CLINICAL TRIAL: NCT06248203
Title: Teachers Delivering Task-Shifted Mental Health Care to Adolescents in India
Brief Title: Teachers Leading the Front Lines - Adolescent
Acronym: TeaLeaf-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of North Bengal, India (Unknown); Darjeeling Ladenla Road Prerna (Unknown); Broadleaf Health and Education Alliance (Other); University of Colorado, Denver (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-1838
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Behavior; Adolescent - Emotional Problem; Mental Health Issue; Psychosocial Functioning; Depression; Anxiety
MeSH Terms: conditions — Adolescent Behavior; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a non-randomized cluster-controlled pre-post study. Given the nature of the intervention, each school will be a cluster. All schools will initially receive the control condition (EUC) and will be transitioned into the intervention arm (Tealeaf). A qualitative exploration of context and process will be embedded within the framework of the study. An embedded approach has been chosen to facilitate a high level of integration between the qualitative and quantitative components of the study.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded; adolescents must assent, and parents consent, to receive mental health care and teachers will be aware they are delivering care. One research assistant (RA) will not be blinded to observe teachers' fidelity. Otherwise, personnel are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tealeaf - Adolescent (Experimental): The Tealeaf-A arm will have three randomized schools. Teachers in the Tealeaf-A arm will receive six days of training and then supervision every 2 weeks to deliver care.
  Interventions: Behavioral: Tealeaf-Mansik Swasta (Tealeaf) as adapted for Adolescents
- Enhanced Usual Care (EUC) (Active Comparator): The EUC arm will have three randomized schools and will be used as an ethical comparator for the Tealeaf-A arm. Teachers will receive two days of training, all materials, and no supervision.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Tealeaf-Mansik Swasta (Tealeaf) as adapted for Adolescents — The investigators will test Tealeaf (Teachers Leading the Frontlines - Mansik Swastha [Mental Health in Nepali]) as adapted for adolescents. Tealeaf is a task-shifting intervention in which teachers deliver transdiagnostic mental health care. Created in Darjeeling, Tealeaf centers on training and supervising teachers to deliver "education as mental health therapy" (Ed-MH) to children (age 5-12). Ed-MH is the investigators' novel, task-shifting, therapy modality that minimizes the time teachers need to deliver care by fitting it into their work. In Ed-MH, teachers use evidence-based therapeutic techniques adapted for use in their existing interactions with students in need (e.g., while teaching) and streamlined for care for any diagnosis ("transdiagnostic"). Tealeaf-A's adaptation (inclusive of Ed-MH) is supported by a Doris Duke Charitable Foundation (DDCF), Fund to Retain Clinical Scientists (FRCS), Caregivers at Carolina COVID award.
  Other Names: Tealeaf-A
  Arms: Tealeaf - Adolescent
Behavioral: Enhanced Usual Care (EUC) — Enhanced Usual Care (EUC) is a less intensive version of the Tealeaf intervention. The EUC service package has been designed to be the most intensive form of care that could be envisioned as viable in the study setting in the foreseeable future without a significant increase in resource investment.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
Purpose: The purpose of this research is to pilot test a novel, alternative, potentially sustainable system of teacher-delivered, task-shifted adolescent mental health care.

Participants: Principals of 60 rural, low-cost private secondary schools of the Darjeeling Himalayas will be invited to participate as a school and an individual. Teachers will be approached individually. Two students per teacher who meet inclusion criteria will be randomly chosen for enrollment.

Procedures: This is a RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) guided, mixed methods CRCT, clustered at schools, of Tealeaf-A's Reach, Adoption & Implementation (Primary Outcomes, implementation-based), as well as evaluating for preliminary indicators of Effectiveness & Maintenance (Secondary Outcomes, clinically-based).

DETAILED DESCRIPTION:
The overarching goal of this proposal is to address the youth mental health crisis by increasing access to high quality, alternative, sustainable adolescent mental health care. The overall objective of this proposal is to pilot test a novel, alternative, potentially sustainable system of teacher-delivered, task-shifted adolescent mental health care. In Darjeeling, India, the investigators will test Tealeaf (Teachers Leading the Frontlines - Mansik Swastha [Mental Health in Nepali]) as adapted for adolescents (Tealeaf-Adolescent; "Tealeaf-A"). Created in Darjeeling, Tealeaf centers on training and supervising elementary school teachers to deliver "education as mental health therapy" (Ed-MH) to children (age 5-12). Ed-MH is the investigators' novel, task-shifting, therapy modality that minimizes the time teachers need to deliver care by fitting it into their work.8 In Ed-MH, teachers use evidence-based therapeutic techniques adapted for use in their existing interactions with students in need (e.g., while teaching) and streamlined for care for any diagnosis ("transdiagnostic"). Tealeaf-A's adaptation (inclusive of Ed-MH) is supported by a Doris Duke Charitable Foundation (DDCF), Fund to Retain Clinical

Scientists (FRCS), Caregivers at Carolina COVID (Corona Virus Disease) award. The investigators' central hypotheses are that teachers can deliver Tealeaf-A (task-shifted mental health care fitted into their work) with fidelity, stakeholders (teachers, adolescents, parents, principals) will find Tealeaf-A acceptable & feasible, and adolescents in Tealeaf-A will show preliminary indicators of mental health symptom improvement versus a comparator. The investigators' rationale stems from two trials in Darjeeling where mental health symptoms of children in Tealeaf improved from clinical to neurotypical. The investigators propose a mixed methods explanatory sequential study, collecting quantitative (QUAN) then qualitative data (qual) to explain QUAN (QUAN-qual). The investigators' specific aims are:

1. To determine if teachers can deliver Tealeaf-A with fidelity, with positive acceptability & feasibility for stakeholders, and leading to preliminary indicators of improved adolescent mental health outcomes (QUAN). Guided by the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework, the investigators hypothesize that a pilot cluster randomized controlled trial (CRCT) of Tealeaf-A clustered at the school level (n=6 schools, 72 teachers, 144 students) will show that:

   * Hypothesis 1a (H1a): Teachers can deliver Tealeaf-A with fidelity and positive feasibility & acceptability for stakeholders (Reach, Adoption, Implementation; Primary Outcomes), and
   * Hypothesis 1b (H1b): Adolescents in Tealeaf-A will have preliminary indicators of improved student mental health symptoms versus a comparator (Effectiveness, Maintenance; Secondary Outcomes).
2. To explore under what circumstances teachers can deliver Tealeaf-A with fidelity, with positive acceptability & feasibility for stakeholders, and that leads to preliminary indicators of improved adolescent mental health outcomes (qual; QUAN - qual). Guided by the Consolidated Framework for Implementation Research (CFIR), the investigators will explore the role of intervention and contextual factors in Aim 1 outcomes by completing key informant interviews with randomly selected stakeholders stratified by stakeholder group, school, and trial arm (n=42) 3 months Post intervention. Mixed methods data integration will occur in side-by-side QUAN-qual joint display tables. As this Aim is exploratory, it does not have a hypothesis to test. Based on previous results and review of the literature, though, the investigators discuss in Aim 2 in "Research Design & Methods" the anticipated findings.

Tealeaf-A Adaptation:

Implemented over a school year, Tealeaf has six components. (1) Teachers first complete six days of training on components 2-6, delivered by the investigators' local collaborator's team (DLRP) of psychiatric social workers with 8 years of experience with Tealeaf. (2) Teachers then nominate students for care based on their judgment, grounded in their everyday interactions with students. This method was chosen based on accuracy (as in "Evidence") and to avoid 1:1 screenings that may identify to others which students need mental health support. (3) They next analyze these students' symptoms with basic functional behavioral assessments. (4) Informed by behavior analyses, they then develop an individualized response using the 4Cs plan (Cause, Change, Connect, and Cultivate). Behavior plans (4Cs) are the chosen care framework (not manualized care) as they align with how teachers individualize teaching to students' needs. The goal of the 4Cs is to improve mental health through and in addition to learning, whereas typical behavior plans solely target improved learning. Teachers have improved learning but not mental health symptoms when individualizing pedagogy using behavior plans; individualization alone was not sufficient. In the 4Cs, teachers pick transdiagnostic therapeutic techniques to deliver from an Ed-MH menu of evidence-based options. For children, Tealeaf's current target, Ed-MH adapts Cognitive Behavior Play Therapy (CBPT) measures for classroom delivery. Based in Cognitive Behavior Therapy (CBT), CBPT is accessible to children <10 years old using both talk and play therapy. Play therapy for children and CBT for youth >10 years old have repeatedly improved symptoms. Ed-MH techniques include managing behaviors in class, 1:1 sessions, and adjusting knowledge transfer processes. (5) Working with caregivers as they see fit, as professional clinicians do, teachers encourage 4Cs use at home. (6) Teachers deliver Ed-MH over a school year, with supervision every two weeks and guided by iterative 4Cs as students' needs evolve.

The investigators adapted Tealeaf to address adolescent needs (Tealeaf-A) in 2022 with support from a DDCF FRCS award. Adaptations to better target adolescents include: (1) changing Ed-MH techniques from CBPT to CBT (i.e., abstract cognitive concepts rather than play approaches); (2) modifying Tealeaf's structure as students have different teachers for different subjects (where 1 teacher will be the lead and coordinate with other teachers); (3) newly compensating teachers given this additional coordination and for caring for more students since each teacher sees more students as subject teachers; and (4) enhancing confidentiality. Confidentiality adaptations included: (4a) focusing Ed-MH techniques on homework changes rather than classwork to avoid in-class additional attention; (4b) limiting what is shared with caregivers to safety information; and (4c) having discrete spaces in schools to meet 1:1.

Tealeaf and Ed-MH's mechanism of action for improving mental health symptoms is through teachers guiding adolescents to consistently practice coping skills and emotion regulation for long periods of time (a school day) and in real time (in the moments of concern). Like counselors, Tealeaf teachers help students gain insight and acquire coping skills. Teachers take the therapy activities farther, though, by overseeing adolescents practicing coping skills, reinforcing positive behavior, and supporting them in moments of struggle, all in real time. It is ideally how teachers would work with students as guided by a therapist, but here themselves determine how to therapeutically respond to a student's mental health needs since therapists are rare. Moreover, as a role model, teachers already play a key role in the social, emotional, and academic development of students and interact with them individually in moments of concern. Ed-MH allows teachers to deliver therapy in shared moments, in real-time. Professional and lay counselors, instead, can only reflect from afar on moments the student is willing to share in the office.

A second mechanism of action is through teachers delivering care that can target education symptoms of mental health as seen in India. In the Ed-MH example in "Background", the student had poor schoolwork due to anxiety. His teacher can target his poor schoolwork (the education symptom of his mental health) and anxiety by improving schoolwork quality (an education intervention) through building his capacity to complete assignments gradually, i.e., exposure therapy (an evidence-based therapy technique). After care, both symptoms improved.

Intervention evidence: Results from 2018 and 2019 pilot Tealeaf trials show that mental health care delivery for children can be shifted to teachers. (1) Teachers (n=19) nominated students (n=36) with moderate accuracy, 72% sensitivity and 62% specificity, aligned with identification by lay counselors in LMICs (Low- or Middle-Income Countries) and teachers in HICs (High-Income Countries). (2) Teachers (n=19) delivered care with fidelity, on average at or above 60% fidelity to protocol, similar to mental health professionals' fidelity to new therapies. (3) Teachers (n=19) found it feasible to deliver therapy when integrated into their workflow (Ed-MH), citing choice of therapeutic techniques and the ability to incorporate them into teaching.(4) Teachers, families, and students found it acceptable for teachers to deliver mental health care.Teachers cited flexible care delivery, families cited impact, and students cited being treated well. (5) Children's mental health symptoms improved after receiving Ed-MH from their teachers, an early signal of impact. Symptoms improved on average from clinical to neurotypical, i.e., from the 77th to the 60th percentile baseline to end line on a gold standard measure in 2018 (n=36) and from the 84th to the 68th percentile in 2019 (n=26). While supported children in 2019 had neurotypical symptom levels at end line, children receiving enhanced usual care (n=188) remained at clinical levels (81st percentile). These findings support teachers' delivery of task-shifted, indicated child mental health care that is transdiagnostic and integrated into their work. This structure is similar to teacher-delivered adolescent promotion and prevention that has improved mental health outcomes. Thus, a next logical step is to test teachers' delivery of indicated adolescent care structured similarly to (1) adolescent prevention & promotion and (2) indicated children's care.

The investigators' rationale for pilot testing Tealeaf-A is based on Tealeaf's promising results as there is an urgent need to identify and deliver evidence-based adolescent mental health interventions to tackle the adolescent mental health care gap that worsened into a crisis during the COVID pandemic. Adapting Tealeaf to adolescents and its testing would occur ideally after completing the investigators' Type 1 hybrid effectiveness-implementation trial of Tealeaf for children (ongoing, in year 2 of 4). Of note, Tealeaf skipped over efficacy (lab-like setting) to effectiveness testing (real world), as literature supports skipping efficacy testing of task-shifted mental health care. Task-shifting improves mental health outcomes in lab-like settings and is now recommended to be tested in specific forms (e.g., teacher-delivery) for specific contexts to study its effects in real world practice. The high risk of poor care access, such as disability, to a large population of adolescents justifies Tealeaf's accelerated testing based on its promise. Also, recent implementation science literature supports parallel trials of the same intervention to accelerate research translation into practice since evidence takes 17 years on average to reach clinical practice. Supported by literature, creating Tealeaf-A given promising results was then supported by a DDCF FRCS award, further substantiating the accelerated pursuit of Tealeaf-A. Also, Tealeaf-A care delivery would ideally include teachers and peers. Due to resource limitations and prioritizing indicated over complementary care, a teacher-led Tealeaf-A adaptation was prioritized. A grant is pending to develop a peer component.

ELIGIBILITY:
Inclusion Criteria:

Schools:

* LCP (Low-Cost Private) Secondary Schools
* Enrolled families earning <$10 daily
* Located in greater Darjeeling
* Principal must also be eligible to participate

Principals:

* >18 years old
* Employed at enrolled school
* Not suspected or convicted of child maltreatment

Teachers:

* >18 years old
* Employed at enrolled school
* Not suspected or convicted of child maltreatment

Students:

* Age 13 - 17 years
* Student of enrolled teacher
* Borderline or clinical Total Problem or subscale score of YSR (Youth Self-Report) and TRF (Teacher's Report Form)
* Each student has a lead teacher (2/teacher), with their other teachers also involved

Guardians

* >18 years old
* Guardian of enrolled student
* Not suspected or convicted of child maltreatment

Exclusion Criteria:

* Exclusion criteria will be set as each participant not meeting inclusion criteria as set for their group.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Mean Number of Dropouts (Reach) | Month 9 of Academic Years 1 and 2
  Dropout standards were set to indicate positive retention within arm per the investigators' previous trials and CRCTs clustered at schools and between arm per mental health therapy RCTs. Data will be analyzed at month 9 of Academic Years 1 and 2 (with month 0 being the start of training) with means compared to 10% dropout standard within arm.
Applied Mental Health Research Dissemination and Implementation Adoption Scale scores (Adoption) | Month 0, Month 9 of Academic Years 1 and 2
  Each student, guardian, teacher, and principal will fill out the Applied Mental Health Research (AMHR) Dissemination and Implementation (D&I) Adoption scale. In other LMICs, these scales had adequate internal consistencies (0.61 to 0.95). They will be translated into Nepali, back-translated, and reviewed by a study collaborator. Each scale has 13-20 items. Each item is rated from 0 ("not at all") to 3 ("a lot") or "don't know/not applicable"; an average score of 2 or more per scale is a positive outcome.
  Data will be collected at Month 0 (post-training, pre-care) and/or starting at Month 9 (post) of Academic Years 1 and 2
Applied Mental Health Research Dissemination and Implementation Adoption Scale scores (Implementation) | Month 9 of Academic Years 1 and 2
  (3A) Fidelity: Observation checklists are from a 2018 fidelity study. The threshold was set within arm per the 2018 study and between arm per mental health care fidelity RCTs. Data will be collected at Month 9, when teachers are expected to have optimal fidelity across arms. (3B) Feasibility & acceptability: AMHR specifics, data collection timing, and 3A & 3B analyses are per "Adoption".

SECONDARY OUTCOMES:
Change in Teacher's Report Form & Youth Self-Report (Effectiveness) | Month 0 up until Month 21 relative to Academic Years 1 and 2
  To estimate effect sizes for all TRF (Teacher's Report Form) and YSR (Youth Self-Report) scores Pre-Post within arm, and between arms, the investigators will calculate Cohen's d. The TRF measures problem behaviors that children may present in school. This is done through questions about the child's academic performance, questions comparing the child to their peers, and a 112 item scale with answer options from 0 ("not true") to 2 ("very true or often true"). The YSR is a 112 item scale that measures "problem behaviors" with answer options from 0 ("not true") to 3 ("very true or often true"). The investigators will compare scores at these same time points using multilevel, multivariable generalized linear regression models (up to 2 levels [teacher, school]) to (1) account for nested data collection (e.g., 1 teacher rating multiple students) and (2) control for sex/gender, other relevant demographics (e.g., income), and potential confounders (e.g., outpatient care).
Maintenance (Teacher's Report Form & Youth Self-Report) | Month 9, 12, 15, and 21 of Academic Year 2
  For Maintenance, the investigators will compare TRF and YSR scores at Month 9 minus scores at Months 12, 15, and 21 of Academic Year 2 using multilevel, multivariable generalized linear regression models (see "Effectiveness").

CONTACTS AND LOCATIONS:
Overall Officials: Christina Cruz, MD; EdM, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Darjeeling Ladenla Road Prerna, Darjeeling, West Bengal, India

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 12 months after the conclusion of the trial to allow researchers to analyze data and submit for peer review.
Access Criteria: Data will be deposited in UNC Odum Institute's UNC Dataverse, a data repository service for the University of North Carolina at Chapel Hill (UNC) research community and its partners.
URL: https://dataverse.unc.edu

REFERENCES:
- [Background] van Ginneken N, Tharyan P, Lewin S, Rao GN, Meera SM, Pian J, Chandrashekar S, Patel V. Non-specialist health worker interventions for the care of mental, neurological and substance-abuse disorders in low- and middle-income countries. Cochrane Database Syst Rev. 2013 Nov 19;(11):CD009149. doi: 10.1002/14651858.CD009149.pub2. PMID 24249541
- [Background] van Ginneken N, Chin WY, Lim YC, Ussif A, Singh R, Shahmalak U, Purgato M, Rojas-Garcia A, Uphoff E, McMullen S, Foss HS, Thapa Pachya A, Rashidian L, Borghesani A, Henschke N, Chong LY, Lewin S. Primary-level worker interventions for the care of people living with mental disorders and distress in low- and middle-income countries. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD009149. doi: 10.1002/14651858.CD009149.pub3. PMID 34352116
- [Background] Patel V, Kieling C, Maulik PK, Divan G. Improving access to care for children with mental disorders: a global perspective. Arch Dis Child. 2013 May;98(5):323-7. doi: 10.1136/archdischild-2012-302079. Epub 2013 Mar 9. PMID 23476001
- [Background] Shinde S, Weiss HA, Varghese B, Khandeparkar P, Pereira B, Sharma A, Gupta R, Ross DA, Patton G, Patel V. Promoting school climate and health outcomes with the SEHER multi-component secondary school intervention in Bihar, India: a cluster-randomised controlled trial. Lancet. 2018 Dec 8;392(10163):2465-2477. doi: 10.1016/S0140-6736(18)31615-5. Epub 2018 Nov 22. PMID 30473365
- [Background] Burns BJ, Costello EJ, Angold A, Tweed D, Stangl D, Farmer EM, Erkanli A. Children's mental health service use across service sectors. Health Aff (Millwood). 1995 Fall;14(3):147-59. doi: 10.1377/hlthaff.14.3.147. PMID 7498888
- [Background] Kola L, Kohrt BA, Hanlon C, Naslund JA, Sikander S, Balaji M, Benjet C, Cheung EYL, Eaton J, Gonsalves P, Hailemariam M, Luitel NP, Machado DB, Misganaw E, Omigbodun O, Roberts T, Salisbury TT, Shidhaye R, Sunkel C, Ugo V, van Rensburg AJ, Gureje O, Pathare S, Saxena S, Thornicroft G, Patel V. COVID-19 mental health impact and responses in low-income and middle-income countries: reimagining global mental health. Lancet Psychiatry. 2021 Jun;8(6):535-550. doi: 10.1016/S2215-0366(21)00025-0. Epub 2021 Feb 24. PMID 33639109
- [Background] Liang L, Ren H, Cao R, Hu Y, Qin Z, Li C, Mei S. The Effect of COVID-19 on Youth Mental Health. Psychiatr Q. 2020 Sep;91(3):841-852. doi: 10.1007/s11126-020-09744-3. PMID 32319041
- [Background] Frontiers Production Office. Erratum: The Potential Emergence of "Education as Mental Health Therapy" as a Feasible Form of Teacher-Delivered Child Mental Health Care in a Low and Middle Income Country: A Mixed Methods Pragmatic Pilot Study. Front Psychiatry. 2022 Jan 18;12:838044. doi: 10.3389/fpsyt.2021.838044. eCollection 2021. PMID 35115975
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Wong G, Greenhalgh T, Westhorp G, Buckingham J, Pawson R. RAMESES publication standards: realist syntheses. J Adv Nurs. 2013 May;69(5):1005-22. doi: 10.1111/jan.12095. Epub 2013 Jan 29. PMID 23356726
- [Background] Pawson R, Greenhalgh T, Harvey G, Walshe K. Realist review--a new method of systematic review designed for complex policy interventions. J Health Serv Res Policy. 2005 Jul;10 Suppl 1:21-34. doi: 10.1258/1355819054308530. PMID 16053581
- [Background] Cruz CM, Dukpa C, Vanderburg JL, Rauniyar AK, Giri P, Bhattarai S, Thapa A, Hampanda K, Gaynes BN, Lamb MM, Matergia M. Teacher, caregiver, and student acceptability of teachers delivering task-shifted mental health care to students in Darjeeling, India: a mixed methods pilot study. Discov Ment Health. 2022;2(1):21. doi: 10.1007/s44192-022-00024-z. Epub 2022 Oct 31. PMID 36341156
- [Background] Pearson N, Naylor PJ, Ashe MC, Fernandez M, Yoong SL, Wolfenden L. Guidance for conducting feasibility and pilot studies for implementation trials. Pilot Feasibility Stud. 2020 Oct 31;6(1):167. doi: 10.1186/s40814-020-00634-w. PMID 33292770
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272